CLINICAL TRIAL: NCT06570564
Title: Upper Versus Lower Limb Exercises on Intermittent Claudication in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, El-Sayed Essam, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16122022
Record Dates: First submitted 2024-04-18; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-04

CONDITIONS: Intermittent Claudication
MeSH Terms: conditions — Intermittent Claudication | interventions — Exercise Test

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Upper limb exercises group. (Experimental): Upper limb exercises group consist of 20 patients. They received arm cranking exercise and routine physiotherapy program.
  Interventions: Device: The arm crank ergometer; Device: treadmill
- Lower limb exercises group. (Experimental): Lower limb exercises group consist of 20 patients. They received bicycling exercise and routine physiotherapy program.
  Interventions: Device: bicycle ergometer; Device: treadmill
- The control group. (Experimental): The control group consisted of 20 patients. They received only routine physiotherapy program.
  Interventions: Device: treadmill

INTERVENTIONS:
Device: The arm crank ergometer — Before starting the program, patients will perform an adaptation session for familiarization with the ergometer and also to identify the training load. For this, patients will perform 10 bouts of two minutes of exercising with a minimum load and two minute passive intervals between bouts. Patients will be instructed to maintain 50 revolutions per minute (RPM) during the exercise. Subsequently, to determine the training load for each session, patients will perform a progressive test where the load will be increased by 10 watts every minute of the test, following the protocol of two minutes of exercise with two minutes of interval
  Arms: Upper limb exercises group.
Device: bicycle ergometer — bicycle ergometer program will consist of a bicycling exercise 3 days per week. Exercise intensity was set at 70% of maximal load with 30 minutes per session. The exercise protocol also incorporated warm-up and cool-down sessions that involved stretches of the major lower limb muscle groups (total exercise time, 40-60 minutes)
  Arms: Lower limb exercises group.
Device: treadmill — Supervised treadmill exercise as routine physiotherapy program

SUMMARY:
Sixty patients with intermittent claudication and type 2 diabetes mellitus. Their age will ranged from 45-55 years old. They recruited from internal department at Damanhour Medical National Institute (DMNI), Damanhour, Beheira Governorate, Egypt. Patients randomly assigned into three equal groups:

Group (A):

Upper limb exercises group consist of 20 patients. They received arm cranking exercise three times per week for three consecutive months plus routine physiotherapy program.

Group (B):

Lower limb exercises group consist of 20 patients. They received bicycling exercise three times per week for three consecutive months plus routine physiotherapy program.

Group (C):

The control group consisted of 20 patients. They received only routine physiotherapy program.

DETAILED DESCRIPTION:
1. Subjects:

   Sixty patients with intermittent claudication and type 2 diabetes mellitus. Their age ranged from 45-55 years old. They recruited from internal department at Damanhour Medical National Institute (DMNI), Damanhour, Beheira Governorate, Egypt. Patients randomly assigned into three equal groups:

   Group (A):

   Upper limb exercises group consist of 20 patients. They received arm cranking exercise three times per week for three consecutive months plus routine physiotherapy program.

   Group (B):

   Lower limb exercises group consist of 20 patients. They received bicycling exercise three times per week for three consecutive months plus routine physiotherapy program.

   Group (C):

   The control group consisted of 20 patients. They received only routine physiotherapy program.
2. Equipment:

Measurement equipment:

1. The Treadmill:

   All patients were tested Maximum walking distance and Pain free walking distance by walking in the treadmill.
2. Ankle/brachial indices (ABI) Doppler Ultrasound Machine
3. All patients were tested HbA1C before and after the treatment in medical analysis lab department at Damanhour Medical National Institute (DMNI).

Therapeutic equipment:

1. The arm crank ergometer
2. bicycle ergometer

ELIGIBILITY:
Inclusion Criteria:

* Sixty patients with type 2 diabetes mellitus and intermittent claudication.
* Patients with diabetes at least 5 years.
* Both genders were included.
* Their age will be ranged from 45-55 years old.
* Patients referred from physician of internal medicine diagnosed as controlled type 2 diabetes (HbA1c 7-7.5%) for the previous 3 months.
* Their body mass index will be ranged from 25.0 to 34.9 kg/m2.

Exclusion Criteria:

* Pregnant women.
* Malignancy.
* Other medical conditions such as uncontrolled hypertension and osteoporosis.
* Past medical history included conditions that may influence the provision of physiotherapy interventions such as (severe asthma, chronic airflow limitation, bronchiectasis, ankylosing spondylitis or lumbar disc prolapse).

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
maximum walking distance (MWD) in meter | three consecutive months
  the distance that had been walked on the treadmill when patients were unable to continue because of severe claudication pain
pain free walking distance (PFWD) in meter | three consecutive months
  the distance that patients can walk on the treadmill before claudication pain begins
claudication score | three consecutive months
  Claudication pain scale is a continuous scale from 1, indicating no pain, to 5 indicating severe pain
Ankle/brachial indices (ABI) by doppler ultrasound | three consecutive months
glycated haemoglobin (HbA1C) | three consecutive months
  It is the average of blood glucose (sugar) levels for the last two to three months. If you have diabetes, an ideal HbA1c level is 48mmol/mol (6.5%) or below

CONTACTS AND LOCATIONS:
Locations (1):
- Damanhour teaching hospital, Damanhūr, Damanhour, Egypt

IPD SHARING:
Plan to Share IPD: No